CLINICAL TRIAL: NCT03607279
Title: Comparison of Plasma Neutrophil Gelatinase - Associated Lipocalin (NGAL) Levels After Robot-assisted Laparoscopic Versus Retropubic Radical Prostatectomy
Brief Title: Comparison of Plasma Neutrophil Gelatinase - Associated Lipocalin (NGAL) Levels
Status: Completed | Type: Observational
Sponsor: Antalya Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Arzu Karaveli, Study director, Antalya Training and Research Hospital
Other Study IDs: 2016-118
Record Dates: First submitted 2018-07-23; First posted 2018-07-31 (Actual); Last update posted 2018-12-19 (Actual); Status verified 2018-12

CONDITIONS: Prostatectomy
Keywords: NGAL; Prostatectomy; Acute kidney injury
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- NGAL - retropubic radical prostatectomy: Plasma NGAL was determined at baseline, 6 and 12 hrs after induction of anaesthesia
  Interventions: Procedure: NGAL
- NGAL - robotic radical prostatectomy: Plasma NGAL was determined at baseline, 6 and 12 hrs after induction of anaesthesia
  Interventions: Procedure: NGAL

INTERVENTIONS:
Procedure: NGAL

SUMMARY:
The purpose of the study is to compare the effect of two surgical techniques (open vs robotic assisted) on plasma levels of NGAL (neutrophil gelatinase-associated lipocalin) after radical prostatectomy.

DETAILED DESCRIPTION:
Patients undergoing radical prostatectomy are at increased risk of acute kidney injury (AKI) because of intraoperative bleeding, obstructive uropathy and older age. In particular robot-assisted laparoscopic radical prostatectomy (RALP) which is in increasing demand as an alternative surgical option for retropubic radical prostatectomy (RRP) is associated with postoperative renal dysfunction because pneumoperitoneum during RALP can decrease cardiac output and renal perfusion. NGAL may become important for diagnosis of postoperative AKI after urogenital oncosurgery.

ELIGIBILITY:
Inclusion Criteria:

* patients who undergo prostatectomy
* American Society of Anesthesiology (ASA) I-III

Exclusion Criteria:

* preexisting renal disease
* emergency surgery
* heart failure
* peripheral vascular disease

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: prostatectomy
Sampling Method: Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Plasma NGAL | 0 hours, 6 hours and 12 hours after surgery
  Plasma NGAL was determined at baseline, 6 hours and 12 hours after surgery, ng/ml

CONTACTS AND LOCATIONS:
Overall Officials: Arzu Karaveli, Principal Investigator — Netherlands: Ministry of Health, Welfare and Sports
Locations (1):
- Antalya Training and Research Hospital, Department of Anesthesiology and Reanimation, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Orsolya M, Attila-Zoltan M, Gherman V, Zaharie F, Bolboaca S, Chira C, Bodolea C, Tomuleasa C, Irimie A, Coman I, Ionescu D. The effect of anaesthetic management on neutrophil gelatinase associated lipocalin (NGAL) levels after robotic surgical oncology. J BUON. 2015 Jan-Feb;20(1):317-24. PMID 25778333
- [Background] Joo EY, Moon YJ, Yoon SH, Chin JH, Hwang JH, Kim YK. Comparison of Acute Kidney Injury After Robot-Assisted Laparoscopic Radical Prostatectomy Versus Retropubic Radical Prostatectomy: A Propensity Score Matching Analysis. Medicine (Baltimore). 2016 Feb;95(5):e2650. doi: 10.1097/MD.0000000000002650. PMID 26844486